CLINICAL TRIAL: NCT01083342
Title: Open-labeled, Multicenter Phase II Study of High-Dose (HD) Methotrexate (MTX) Induction Chemotherapy Followed by Alternative HD MTX-based and HD Cytarabine-based Combination Consolidation Chemotherapy for Newly Diagnosed Primary CNS Lymphoma; CISL 10-01 Study
Brief Title: High-Dose (HD) Methotrexate (MTX) Induction Chemotherapy Followed by Alternative HD MTX-based and HD Cytarabine-based Combination Consolidation Chemotherapy for Newly Diagnosed Primary CNS Lymphoma; CISL 10-01 Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-12-087
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: CNS Lymphoma
Keywords: primary CNS lymphoma; MTX: Methotrexate,Leucovorin; MVD: Methotrexate,Vincristine,Dexamethasone; VIA: VP-16 (Etoposide),Ifosfamide,Mesna, Cytarabine (ara-C); Newly diagnosed primary CNS lymphoma patients

INTERVENTIONS:
Drug: MTX, MVD, VIA — MTX: Methotrexate,Leucovorin MVD: Methotrexate,Vincristine,Dexamethasone VIA: VP-16 (Etoposide),Ifosfamide,Mesna, Cytarabine (ara-C)

SUMMARY:
The purpose of this study is to evaluate the complete response (CR) rate after HD-MTX induction chemotherapy followed by alternative HD MTX-based and HD Cytarabine-based combination consolidation chemotherapy

ELIGIBILITY:
Inclusion criteria

1. Histologically confirmed Primary Central Nervous System (CNS) lymphoma
2. Previously untreated. Patients treated with steroid alone are eligible.
3. Performance status: ECOG 0-3.
4. Age; 20-70
5. Adequate renal function: Estimated glomerular filtration rate (GFR) or estimated creatinine clearance (CrCl) ≥ 50 mL/min
6. Adequate liver functions: Transaminase (AST/ALT) < 3 X upper normal value & Bilirubin < 2 X upper normal value
7. Adequate hematological function: hemoglobin ≥ 9 g/dL absolute neutrophil count (ANC) ≥ 1,500/μL and platelet count ≥ 75,000/μL
8. At least one cerebral mass lesion on magnetic resonance imaging (MRI) without involvement beyond the central nervous system (CNS)
9. Life expectancy > 6 months
10. A negative serum or urine pregnancy test prior to treatment must be available both for pre menopausal women and for women who are < 1 years after the onset of menopause.
11. Informed consent

Exclusion criteria

1. Other subtypes NHL than Primary Central Nervous System (CNS) lymphoma
2. Systemic involvement of Primary CNS lymphoma except leptomeningeal involvement
3. Intraocular lymphoma
4. HIV (+)
5. Any other malignancies within the past 5 years except curatively treated non-melanoma skin cancer or in situ carcinoma of cervix uteri
6. Pregnant or lactating women, women of childbearing potential not employing adequate contraception
7. Other serious illness or medical conditions

   * Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry
   * History of significant neurological or psychiatric disorders
   * Active uncontrolled infection (viral, bacterial or fungal infection)
8. Patients who have HBV (+) are eligible. However, primary prophylaxis using antiviral agents (i.e. lamivudine) is recommended for HBV carrier to prevent HBV reactivation during whole treatment period.
9. Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the complete response (CR) after chemotherapy | 24 months

SECONDARY OUTCOMES:
To evaluate the duration of response | 24 months
To evaluate the progression-free survival, overall survival | 24 months
To evaluate the safety profiles | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: WonSeog Kim,, M.D., PhD., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea